CLINICAL TRIAL: NCT06824350
Title: Multi-component Chlorination Intervention to Reduce Neonatal Infections in Rural Health Facilities
Brief Title: Clean Trial - Chlorination to Reduce Enteric and Antibiotic Resistant Infections in Neonates
Acronym: CLEAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Kenya Medical Research Institute (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-01-17100; R01AI184756 (NIH)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sepsis; Neonatal Mortality; Antibiotic Resistant Infection; Enteric Infections; Serious Bacterial Infection
Keywords: infection prevention and control; antibiotic resistance; bacterial enteric infection; neonatal mortality; sepsis; water disinfection; chlorine; sodium hypochlorite; hospital acquired infections
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Lab technicians will be masked to intervention status of samples received. A subset of investigators will be masked to outcomes by intervention status until data collection is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Control group. At the conclusion of the trial, facilities will receive a chlorine doser.
  Interventions: Behavioral: infection prevention and control messaging
- Multi-component chlorine intervention (Experimental): Health care facilities will receive one or more inline chlorine dosers that will automatically chlorinate all water accessed by the maternity wards. Intervention facilities will also be randomized to either receive an electrochlorinator for on-site production of liquid chlorine solution or to receive bulk chlorine deliveries. Chlorine will be use to refill the chlorine dosers and for surface disinfection. Facilities will also receive hardware to facilitate surface disinfection.
  Interventions: Device: chlorination for water disinfection and surface disinfection; Behavioral: infection prevention and control messaging

INTERVENTIONS:
Device: chlorination for water disinfection and surface disinfection — * Installation of inline chlorine doser(s) for automated water disinfection.
  * Provision of chlorine solution for water and surface disinfection (half of treatment facilities randomized to receive electrochlorinator, half receive bulk chlorine solution deliveries).
  * Provision of mop(s), bucket(s), and spray bottles for surface cleaning.
  Arms: Multi-component chlorine intervention
Behavioral: infection prevention and control messaging — Infection prevention and control guidance and messaging

SUMMARY:
The CLEAN (ChLorine to reduce Enteric and Antibiotic resistant infections in Neonates) cluster randomized controlled trial in western Kenya will evaluate the impact of a multi-component chlorination intervention in health care facilities on maternal and neonatal health. Intervention facilities will receive a passive chlorination technology for water supply treatment and a reliable supply of sodium hypochlorite disinfectant. Both intervention and treatment facilities will receive infection prevention and control messaging. The goal of the study is to evaluate the impact of the intervention on bacterial contamination of water supply, on staff hands, and on high-touch surfaces in maternity wards, and the following outcomes among facility-born neonates and their mothers: (1) gut carriage of bacterial pathogens associated with sepsis one week post-birth, (2) gut carriage of antibiotic resistant bacteria one week post-birth, and (3) symptoms of possible serious bacterial infection one week following birth.

DETAILED DESCRIPTION:
The proportion of births occurring at healthcare facilities is rising globally, yet healthcare facilities in low-income settings have been found to be highly contaminated with bacterial pathogens, including antibiotic resistant pathogens. There is a need for effective strategies to reduce contamination in healthcare facilities in order to reduce infection risks among facility-born neonates. In this trial, medium-sized public health facilities will be randomized to control or to receive an intervention consisting of passive chlorination for water supply treatment and a reliable supply of chlorine disinfectant. Reliable supply is randomized as either (a) an electrochlorinator for on-site production or (b) bulk chlorine delivery.

This cluster randomized controlled trial will enroll 36 health facilities to generate rigorous evidence on the maternal and neonatal health benefits of chlorinated water supply paired with reliable supplies of chlorine disinfectant. This study has the following aims: 1) determine the impact of the intervention on pathogenic and antibiotic resistant bacterial contamination in water supplies, on high-touch surfaces, and on healthcare worker hands, 2) quantify intervention effects on gut colonization of mothers and neonates by a panel of pathogenic and antibiotic resistant bacteria species linked to serious infection, using molecular and culture-based methods, and 3) follow up with mother-neonate dyads to measure intervention effects on symptoms of possible serious bacterial infection in the week following birth. Data collection will be for a duration of 24 months.

Infection prevention through effective water, sanitation, and hygiene (WASH) has been cited by national action plans as a key tool in the fight against antimicrobial resistance and, while global data show dire WASH conditions in low- and middle-income (LMIC) health facilities, there exists very little guidance for implementing effective interventions. The overarching goal is to generate actionable evidence to inform investments in chlorination at health facilities to improve maternal and neonatal health and reduce the threat of antibiotic resistant infections.

ELIGIBILITY:
Facility Inclusion Criteria:

* Public health care facility
* 25 live births or more per month
* Infrastructure compatible with inline chlorination device

Participant Inclusion Criteria:

* Pregnant adults/mature minors arriving at enrolled facilities to give birth and their neonates

Facility Exclusion Criteria:

* Existing facility-level chlorination

Participant Exclusion Criteria:

* Miscarriage (<28 weeks gestation)
* Stillbirth (for neonatal analysis only)
* Unable to give informed consent/do not consent
* Reside >2 hours away from facility for enrollment into swab sampling cohort

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45450 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Possible serious bacterial infection in neonate | From birth to 7 days post birth
  Incidence of one or more of the following severe infection symptoms of neonates based on WHO criteria for possible serious bacterial infection:
  1. Not able to feed at all or not feeding well
  2. Convulsions
  3. Severe chest indrawing
  4. Fever - High body temperature (38°C* or above)
  5. Low body temperature (less than 35.5°C*)
  6. Movement only when stimulated or no movement at all
  7. Fast breathing (60 breaths per minute or more)
Possible maternal sepsis | From birth to 7 days post birth
  Any of the following listed with fever or hypothermia:
  1. fast heartbeat
  2. low blood pressure
  3. respiratory distress
  4. jaundice
  5. decreased urination/dysuria
  6. altered mental status
Neonatal infection with at least one bacterial pathogen | 7 days after birth
  Detection of any pre-specified bacterial pathogen detected by qPCR in infant rectal swabs (among swab subset of participants)
  Includes:
  ETEC, STEC, EPEC, EAEC, EIEC, EHEC O157:H7, Escherichia coli/Shigella, Shigella spp, Shigella flexneri, Salmonella spp., Salmonella enteritidis, Salmonella typhi, Campylobacter jejuni/coli, Staphylococcus aureus, Klebsiella pneumoniae, Streptococcus pneumoniae, Streptococcus agalactiae (Group B strep), Serratia marcescens, Pseudomonas aeruginosa, Acinetobacter baumannii, Clostridium difficile, Vibrio cholerae

SECONDARY OUTCOMES:
Any symptom or sign of infection in neonate | From birth until 7 days post birth
  One or more of the following symptoms:
  Difficulty feeding, Hyperthermia/fever, Hypothermia, Tachypnea, Severe chest indrawing, Convulsions, Movement only when stimulated/no movement, Bulging fontanel, Labored breathing, Skin infection, Umbilical redness, Oozing ears, Diarrhea, Three or more loose or watery stools in a 24 hour period, Vomiting, Cyanosis, Cough, Runny nose or congestion, Tachycardia (>160 bpm at rest)
Any symptom or sign of infection in mother | From birth to 7 days post birth
  One or more of the following symptoms:
  Hypothermia, Fever, Foul smelling vaginal discharge, Fits/convulsions, Tachycardia (>100 bpm at rest), Low blood pressure, Diarrhea (self-defined), Difficulty breathing, Jaundice, Decreased urination or difficult or painful urination, Confusion or altered mental state, Mastitis, Chills, Body aches, Low appetite, Lower abdominal pain, Three or more loose or watery stools in a 24 hour period, Vomiting, Cough, Runny nose or congestion, Chest pain, Bloody stool, Skin infection
Clinical diagnosis of sepsis in neonate | From birth to 7 days post birth
  Abstracted diagnosis from medical charts OR self-reported diagnosis confirmed by clinician
Clinical diagnosis of sepsis in mother | From birth to 7 days post birth
  Abstracted diagnosis from medical charts OR self-reported diagnosis confirmed by clinician
Neonatal mortality | From birth to 28 days after birth
  Report of neonatal death up to 28 days
Maternal mortality | From birth to 28 days after birth
  Report of maternal death
Neonatal rectal colonization with at least one bacterial pathogen by culture | 7 days after birth
  Detection of any pre-specified bacterial pathogen detected by culture in neonate rectal swabs (among swab subset of participants)
  Includes:
  Acinetobacter spp., Pseudomonas spp., Salmonella spp., Shigella, Staphylococcus aureus, Group B streptococcus
Maternal rectal colonization with at least one bacterial pathogen by culture-based method | 7 days postpartum
  Detection of any pre-specified bacterial pathogen detected by culture in maternal rectal swabs (among swab subset of participants)
  Acinetobacter spp., Pseudomonas spp., Salmonella spp., Shigella spp., Staphylococcus aureus, Group B streptococcus
Number of clinically relevant antibiotic resistance genes (ARGs) detected in neonatal rectal swabs | 7 days post birth
  Measured by qPCR. Includes: resistance to quinolone, macrolide, sulfonamide, tetracycline, vancomycin, aminoglycoside, beta-lactams (cephalosporin, penicillin, ampicillin) , carbapenem, colistin
Rectal colonization with one or more antibiotic resistant bacteria (neonates) | 7 days post birth
  Detection of ESBL enterobacteriaceae by culture in rectal swabs
  Includes: Klebsiella spp./Enterobacter/Citrobacter spp. (KEC), Acinetobacter spp., Pseudomonas spp., E. coli
Rectal colonization with one or more antibiotic resistant bacteria (mothers) | 7 days postpartum
  Detection of ESBL enterobacteriaceae by culture in rectal swabs
  Includes: Klebsiella spp./Enterobacter/Citrobacter spp. (KEC), Acinetobacter spp., Pseudomonas spp., E. coli
Number of bacterial pathogens in rectal swabs (neonates) | 7 days post birth
  Number of unique bacterial pathogens (see pre-specified list above) detected by qPCR
Number of bacterial pathogens in rectal swabs (mothers) | 7 days postpartum
  Number of unique bacterial pathogens (see pre-specified list above) by culture

OTHER OUTCOMES:
Rectal colonization with individual bacterial pathogens (neonates) | 7 days post birth
  Detection of individual bacterial pathogen by qPCR or by culture (see list in secondary outcomes)
Rectal colonization with individual bacterial pathogens (mothers) | 7 days postpartum
  Detection of individual bacterial pathogen (see pre-specified list in secondary outcomes) by culture or qPCR
Presence of individual ARGs in neonatal rectal swabs | 7 days post birth
  Presence/absence of pre-specified clinically relevant ARGs by qPCR
Presence and concentration of bacterial pathogens on high touch surfaces | Measured quarterly over 24 months post intervention delivery (every 3 months)
  Measured by culture-based assays
  Includes: Acinetobacter spp., Pseudomonas spp., Salmonella spp., Shigella, Staphylococcus aureus, Group B streptococci
Presence and concentration of antibiotic resistant bacterial pathogens on high touch surfaces | Measured quarterly over 24 months post intervention delivery (every 3 months)
  Detection of ESBL enterobacteriaceae by culture in surface swabs
  Includes: Klebsiella spp./Enterobacter/Citrobacter spp. (KEC), Acinetobacter spp., Pseudomonas spp., E. coli
Proportion of water samples meeting WHO "safe" criteria | Measured quarterly over 24 months post intervention delivery (every 3 months)
  Measured as <1 CFU E. coli per 100ml water tested by culture
Concentration of E. coli / 100 ml water | Measured quarterly over 24 months post intervention delivery (every 3 months)
  Measured by culture-based membrane filtration assay
Presence and concentration of E. coli and total coliform on healthcare staff hands | Measured quarterly over 24 months post intervention delivery (every 3 months)
  Measured by membrane filtration culture assay
Presence and concentration of antibiotic resistant bacterial pathogens on healthcare staff hands | Measured quarterly over 24 months post intervention delivery (every 3 months)
  Detection of ESBL enterobacteriaceae by culture in hand rinses and swabs
  Includes: Klebsiella spp./Enterobacter/Citrobacter spp. (KEC), Acinetobacter spp., Pseudomonas spp., E. coli
Proportion of water supply samples with detectable free chlorine residual in water | Measured quarterly over 24 months post intervention delivery (every 3 months)
  Measured as >0.1 ppm by DPD method

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Pickering, PhD, Principal Investigator — University of California, Berkeley; Phelgona Otieno, PhD, Principal Investigator — Kenya Medical Research Institute; Lillian Musila, PhD, Principal Investigator — Walter Reed Army Institute of Research-Africa
Locations (2):
- University of California, Berkeley, Berkeley, California, United States
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
Any data shared will be de-identified. Participants will not be contacted or re-consented for future sharing or accessing data through repositories. Privacy and confidentiality protections will be consistent with applicable local laws in Kenya. Data will be de-identified prior to sharing. All data sharing plans will be reviewed and approved by the respective institutional review boards at all participating institutions and will be reviewed during the informed consent process with caregivers.

REFERENCES:
- [Background] Lindmark M, Cherukumilli K, Crider YS, Marcenac P, Lozier M, Voth-Gaeddert L, Lantagne DS, Mihelcic JR, Zhang QM, Just C, Pickering AJ. Passive In-Line Chlorination for Drinking Water Disinfection: A Critical Review. Environ Sci Technol. 2022 Jul 5;56(13):9164-9181. doi: 10.1021/acs.est.1c08580. Epub 2022 Jun 14. PMID 35700262
- [Background] Pickering AJ, Crider Y, Sultana S, Swarthout J, Goddard FG, Anjerul Islam S, Sen S, Ayyagari R, Luby SP. Effect of in-line drinking water chlorination at the point of collection on child diarrhoea in urban Bangladesh: a double-blind, cluster-randomised controlled trial. Lancet Glob Health. 2019 Sep;7(9):e1247-e1256. doi: 10.1016/S2214-109X(19)30315-8. PMID 31402005